CLINICAL TRIAL: NCT07026110
Title: Clinical Application Study of PET/CT for Differential Diagnosis of Non-small Cell Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LY2024-329-C
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer; Lung Diseases; Lung Neoplasms; Lung Cancer Metastatic; Lung Inflammation
Keywords: Trophoblast cell surface antigen 2 (Trop2); Epithelial cell adhesion molecule(EpCAM); ImmunoPET; Lung tumor
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases; Pneumonia; Colorectal Cancer, Hereditary Nonpolyposis, Type 8

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ImmunoPET imaging in patients with lung cancers (Experimental): Enrolled lung cancer patients will undergo a Trop2/EpCAM-targeted immunoPET/CT scanning.
  Interventions: Drug: [68Ga]Ga-NOTA-T4; Drug: [68Ga]Ga-NOTA-RT4; Drug: [18F]F-RESCA-T4; Drug: [18F]F-RESCA-RT4; Drug: [18F]F-RESCA-EPCD6; Drug: [68Ga]Ga-NOTA-EPCD6

INTERVENTIONS:
Drug: [68Ga]Ga-NOTA-T4 — Enrolled patients will receive 0.05-0.1 mCi/kg of [68Ga]Ga-NOTA-T4. ImmunoPET/CT imaging will be acquired 1-2 hours after [68Ga]Ga-NOTA-T4 injection.
  Other Names: [68Ga]T4
Drug: [68Ga]Ga-NOTA-RT4 — Enrolled patients will receive 0.05-0.1 mCi/kg of [68Ga]Ga-NOTA-RT4. ImmunoPET/CT imaging will be acquired 1-2 hours after [68Ga]Ga-NOTA-RT4 injection.
  Other Names: [68Ga]RT4
Drug: [18F]F-RESCA-T4 — Enrolled patients will receive 0.05-0.1 mCi/kg of [18F]F-RESCA-T4. ImmunoPET/CT imaging will be acquired 1-2 hours after [18F]F-RESCA-T4 injection.
  Other Names: [18F]T4
Drug: [18F]F-RESCA-RT4 — Enrolled patients will receive 0.05-0.1 mCi/kg of [18F]F-RESCA-RT4. ImmunoPET/CT imaging will be acquired 1-2 hours after [18F]F-RESCA-RT4 injection.
  Other Names: [18F]RT4
Drug: [18F]F-RESCA-EPCD6 — Enrolled patients will receive 0.05-0.1 mCi/kg of [18F]F-RESCA-EPCD6. ImmunoPET/CT imaging will be acquired 1-2 hours after [18F]F-RESCA-EPCD6 injection.
  Other Names: [18F]F-EPCD6
Drug: [68Ga]Ga-NOTA-EPCD6 — Enrolled patients will receive 0.05-0.1 mCi/kg of [68Ga]Ga-NOTA-EPCD6. ImmunoPET/CT imaging will be acquired 1-2 hours after [68Ga]Ga-NOTA-EPCD6 injection.
  Other Names: [18F]F-EPCD6

SUMMARY:
This study aims to explore the efficacy of Trop2, EpCAM-specific PET/CT imaging for noninvasive visualization of Trop2 or EpCAM expression levels in non-small cell lung cancer; and to explore the differences between novel target-specific PET/CT examinations and conventional 18F-FDG PET/CT in the diagnosis and differential diagnosis of solid lung nodules.

DETAILED DESCRIPTION:
A solid lung nodule was initially diagnosed as non-small cell lung cancer by chest CT. Patients with lung nodules subjected to 18F-FDG PET/CT with surgical resection/biopsy. Patients will also be included for routine follow-up, surveillance, and treatment efficacy evaluation.Enrolled patients will undergo whole-body immunoPET/CT scans 1-2 hours after tracer injection (0.05-0.1 mCi/kg). The uptake of imaging tracers in tumors and normal organs/tissues will be scored visually and quantitatively.Tumor uptake will be quantified by the maximum standard uptake value (SUVmax). The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and accuracy will be calculated to assess the diagnostic efficacy. The correlation between lesion uptake and Trop2 and EpCAM expression level determined by immunohistochemistry staining will be further analyzed. The primary exploration endpoint will be the tracers' imaging feasibility and preliminary diagnostic value compared to conventional imaging approaches like 18F-FDG PET/CT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years;
2. Imaging studies suspecting non-small cell lung cancer;
3. Solid lung nodules (≥8 mm in diameter) diagnosed by chest ct, which are subject to 18F-FDG PET/CT and surgical resection/biopsy of lung nodules according to the NCCN guideline specifications for NSCLC in the 2024 edition;
4. Patients or family members agreed to participate in this clinical study and signed an informed consent form.

Exclusion Criteria:

1. Women during pregnancy and lactation;
2. Persons with a history of surgery and trauma that significantly affects metabolic distribution and anatomical structure;
3. Persons with severe other systemic diseases or known hypersensitivity to humanized monoclonal antibody products;
4. Patient is unable to cooperate in completing the PET/CT examination;
5. Patient has participated in other clinical studies within the past year that have resulted in radiation exposures in excess of an effective dose of 50 mSv, in addition to the radiation exposures anticipated from participation in this clinical study;
6. Patient should not participate in this clinical trial in the opinion of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Biodistribution-Standardized uptake value (SUV) of normal tissues and organs. | 1 day from injection of the tracers
  Measurement of the overall biodistribution of the above tracers in normal tissues and organs (bladder (after voiding), background (pelvic fat), blood, brain, salivary and lacrimal glands, lung, liver, spleen, pancreas, small intestine, and kidneys). To calculate the SUV, circular regions of interest were drawn around the area of focally increased uptake in the transaxial slices and automatically fitted to a three-dimensional volume of interest.
SUV of tumors | 1 day from injection of the tracers
  The SUV of the above tracers in the primary and/or metastatic lesions of the included subjects. To calculate the SUV, circular regions of interest were drawn around the area of focally increased uptake in the transaxial slices and automatically fitted to a three-dimensional volume of interest.
Radiation dosimetry of tissues/organs | 1 day from injection of the tracers
  Measurement of absorbed radiation doses (Gy/MBq) to tissues/organs. The following tissues were included: adrenals, brain, breasts, gallbladder, small intestine, upper and lower large intestine, stomach, heart contents, heart muscle, kidney, liver, lung, muscle, ovaries, pancreas, red marrow, trabecular and cortical bone, spleen, testes, thymus, thyroid, urinary bladder, and uterus. Dynamic imaging within one hour will be performed for this purpose.
Radiation dosimetry of tumors | 1 day from injection of the tracers
  Measurement of absorbed radiation doses (Gy/MBq) to tumors. Dynamic imaging within one hour will be performed for this purpose.
Radiation dosimetry of whole-body | 1 day from injection of the tracers
  Whole-body activity was measured using a large volume of interest (VOI) covering the entire subject.
Diagnostic sensitivity | 30 days
  Sensitivity = (True Positives) / (True Positives + False Negatives). The diagnostic value of Trop2 and EpCAM immunoPET/CT will be compared with that of conventional imaging approaches, including 18F-FDG PET/CT, CT, and MRI.
Diagnostic specificity | 30 days
  Specificity = (True Negatives) / (True Negatives + False Positives). The diagnostic value of Trop2 and EpCAM immunoPET/CT will be compared with that of conventional imaging approaches, including 18F-FDG PET/CT, CT, and MRI.
Accuracy | 30 days
  Accuracy = (True Positives + True Negatives) / (Total Tests). The diagnostic value of Trop2 and EpCAM immunoPET/CT will be compared with that of conventional imaging approaches, including 18F-FDG PET/CT, CT, and MRI.
Positive Predictive Value (PPV) | 30 days
  PPV = (True Positives) / (True Positives + False Positives). The diagnostic value of Trop2 and EpCAM immunoPET/CT will be compared with that of conventional imaging approaches, including 18F-FDG PET/CT, CT, and MRI.
Negative Predictive Value (NPV) | 30 days
  NPV = (True Negatives) / (True Negatives + False Negatives). The diagnostic value of Trop2 and EpCAM immunoPET/CT will be compared with that of conventional imaging approaches, including 18F-FDG PET/CT, CT, and MRI.

SECONDARY OUTCOMES:
ImmunoPET/CT in altering initial staging for patients with lung tumors | 3-6 months
  Assess the role of Trop2 and EpCAM immunoPET/CT in initial staging in terms of the number of metastases.
ImmunoPET/CT for postoperative surveillance for patients with lung tumors | 3-6 months
  Assess the role of Trop2 and EpCAMimmunoPET/CT in surveillance in terms of the number of metastases, Trop2 and EpCAM-derived tumor volume (Trop2 and EpCAM-TV), and total lesion Trop2 uptake (Trop2 and EpCAM-TLU).
ImmunoPET/CT for restaging for patients with lung tumors | 3-6 months
  Assess the role of Trop2 and EpCAM immunoPET/CT in restaging in terms of the number of metastases, Trop2 and EpCAM-TV, and Trop2 and EpCAM-TLU.
ImmunoPET/CT in evaluating treatment responses | 1-2years
  We will also investigate the role of Trop2 and immunoPET/CT in predicting and evaluating the treatment efficacy in patients with lung tumors. The treatment regimens involve chemotherapy, molecularly targeted therapies, immunotherapies (e.g. PD-1/PD-L1 inhibitors), and cell therapies.
ImmunoPET/CT in identifying inflammation and tumors in the lungs | 1 day from injection of the tracers
  We will also investigate the role of Trop2 and immunoPET/CT in identifying the benign and malignant nature of pulmonary lesions and hilar and mediastinal lymph nodes

CONTACTS AND LOCATIONS:
Overall Officials: Weijun Wei, Study Chair — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China